CLINICAL TRIAL: NCT04582032
Title: Effects of COX 1-2 Inhibitors on Prevention of Rocuronium Injection Pain: Controlled, Randomised, Double Blind Study
Brief Title: Effects of Cyclooxygenase (COX) 1-2 Inhibitors on Prevention of Rocuronium Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mehmet sahap, Assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: roc
Record Dates: First submitted 2020-09-28; First posted 2020-10-09 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Injection Site Irritation
Keywords: dexketoprofen, pain, rocuronium
MeSH Terms: conditions — Pain | interventions — dexketoprofen trometamol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexketoprofen group, (Active Comparator): IV cannulation was performed on hand dorsum or brachial and canulation place was recorded. Patients allocated in dexketoprofen group were administered intravenous dexketoprofen (50 mg/2ml) and 0,3 mg/kg midazolam 10 minutes prior to general anesthesia induction
  Interventions: Drug: Dexketoprofen (KETAVEL 50 mg/2 ml)
- Saline group (Other): IV cannulation was performed on hand dorsum or brachial and canulation place was recorded. Patients allocated in control group were administered intravenous 2 ml of saline and 0,3 mg/kg midazolam 10 minutes prior to general anesthesia induction
  Interventions: Drug: Saline (Isotonic Saline Solution 0.9% )

INTERVENTIONS:
Drug: Dexketoprofen (KETAVEL 50 mg/2 ml) — intravenous dexketoprofen (KETAVEL 50 mg/2 ml)
  Arms: Dexketoprofen group,
Drug: Saline (Isotonic Saline Solution 0.9% ) — intravenous 2 ml of saline
  Arms: Saline group

SUMMARY:
Purpose : The aim of the study is to investigate the effects of cox inhibitors as a rescue agent against the rocuronium pain Methodology : Sixty patients enrolled for the general anesthesia enrolled in this study. Patients were allocated into two groups (Group 1: Dexketoprofen group, Group 2: Control group) .Pain was evaluated by during rocuronium injection, patients were scored by a scale showed below.

0;No movement response to injection

1. Mild movement response to injection
2. Hand withdrawal response to injection
3. Arm withdrawal response to injection Investigators also evaluated the pain with 2 questions when the patient was in the recovery room.

Question 1.What was the last feeling before participants fall into sleep? question 2. Did participants feel any pain on participants's hand during medication injection for anesthesia?

DETAILED DESCRIPTION:
Purpose : Rocuronium bromide is a painful agent while general anesthesia induction. The aim of the study is to investigate the effects of cox inhibitors as a rescue agent against the rocuronium pain Methodology : Sixty patients enrolled for the general anesthesia enrolled in this study. Patients were allocated into two groups (Group 1: Dexketoprofen group, Group 2: Control group) .Pain was evaluated by during rocuronium injection, patients were scored by a scale showed below.

0;No movement response to injection

1. Mild movement response to injection
2. Hand withdrawal response to injection
3. Arm withdrawal response to injection Investigators also evaluated the pain with 2 questions when the patient was in the recovery room.

Question 1.What was the last feeling before participants fall into sleep? question 2. Did participants feel any pain on participants's hand during medication injection for anesthesia?

ELIGIBILITY:
Inclusion Criteria:

* non allergic to dexketoprofen
* 18-60 years old
* American Society of Anesthesiologists(ASA) 1-2-3
* 70-90 kg weigh

Exclusion Criteria:

* patients with psychiatric and mental problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
The injection pain due to rocuronium | 1 month
  Pain will be recorded and graded using a 4-point scale (none, mild, moderate, or severe).

SECONDARY OUTCOMES:
Score on pain due to injection of rocuronium | 1 month
  Withdrawal reactions are scored as follows: (a) no pain response, (b)pain limited to the wrist, (c) pain limited to the elbow/shoulder, or (d) generalized pain response.

CONTACTS AND LOCATIONS:
Locations (1):
- Kecioren Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No